CLINICAL TRIAL: NCT05787535
Title: A Phase I Study to Evaluate the Safety, Tolerance and Efficacy of HRYZ-T101 TCR-T Cell for HPV18 Positive Advanced Solid Tumor
Brief Title: HRYZ-T101 TCR-T Cell for HPV-18 Positive Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HRYZ Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRYZ-T101-1002
Record Dates: First submitted 2023-03-14; First posted 2023-03-28 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-03

CONDITIONS: Cervical Cancer; Head and Neck Squamous Cell Carcinoma; Oropharyngeal Cancer; Vagina Tumor; Carcinoma of Penis; Anal Carcinoma; Carcinoma of Vulva
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Vaginal Neoplasms; Penile Neoplasms; Anus Neoplasms; Vulvar Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRYZ-T101 TCR-T cell therapy (Experimental): Patients will undergo lymphocytapheresis, then treatment with TCR-T cell.
  Interventions: Drug: Fludarabine + Cyclophosphamide; Biological: HRYZ-T101 TCR-T Cell

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide — Fludarabine: 25mg/m²/day×3days; Cyclophosphamide: 250mg/m²/day×3 days
Biological: HRYZ-T101 TCR-T Cell — On day 1, the TCR-T cells will be administered one time.

SUMMARY:
A single center, open, single arm dose escalation phase I study to evaluate the safety, tolerability, and efficacy of HRYZ-T101 TCR-T cell for HPV18 positive advanced solid tumor. The study will investigate DLT of HRYZ-T101 TCR-T cell injection.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be willing to sign the informed consent form.
2. Age ≥18 years and ≤70 years.
3. Histologically-confirmed advanced metastatic or recurrent solid tumors with confirmed HPV18 infection and HLA-DRB1*09:01 allele.
4. Subjects who have failed at least first-line treatment in the past and lack effective treatment options.
5. ECOG performance status of 0-1.
6. Estimated life expectancy ≥ 3 months.
7. Patients must have at least one measurable lesion defined by RECIST 1.1.
8. Subjects with potential fertility must agree to use effective contraceptive methods during the whole trials period and at least 6 months after receiving HRYZ-T101 cell transfusion treatment.
9. Patients with any organ dysfunction as defined below:

1) Leukocytes≥3.0 x 10^9/L; 2) absolute neutrophil count ≤1.5 x 10^9/L; 3) blood platelets ≥75 x 10^9/L; 4) hemoglobin≥90g/L; 5) Serum albumin ≥ 3.0g/dL; 6) total bilirubin≤1.5×ULN; ALT/AST≤2.5×ULN; 7) Creatinine clearance ≥50mL/min; 8) INR≤1.5×ULN; APTT≤1.5×ULN; 9) LVEF≥50%; 10) SpO2≥92%.

Exclusion Criteria:

1. Organ transplanters and allogeneic cell transplanters.
2. Have a history of hypersensitivity to cyclophosphamide or fludarabine, and it is known that any ingredient used in the treatment of this study will produce allergic reactions.
3. Those who have undergone major surgery within 4 weeks before enrollment, and those who have received conventional chemotherapy, large-area radiotherapy, targeted therapy, endocrine therapy, immunotherapy or biological therapy, and Chinese herbal medicine and other anti-tumor treatment.
4. Have received live attenuated vaccine within 4 weeks before enrollment.
5. Subjects with clinical cardiac symptoms or diseases that cannot be well controlled.
6. The subject has active infection or fever more than 38.5 degrees of unknown cause during screening and before cell transfusion.
7. Subjects have any active autoimmune disease or history of autoimmune disease.
8. Subjects with other malignant tumors.
9. Patients with central nervous system metastasis.
10. Active, uncontrolled bacterial or fungal infection requiring systemic treatment.
11. Known HIV or syphilis infection, and/or active hepatitis B virus or hepatitis C virus infection.
12. It is planned to use immunosuppressive agents, or systemic corticosteroids, immunomodulators.
13. Have received any investigational drug within 4 weeks before enrollment, or have participated in another clinical study at the same time.
14. Pregnant or lactating subjects, or those who are unwilling to contraception during the test.
15. Known uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease or liver failure.
16. Other serious organic diseases and mental disorders.
17. Have received any gene therapy products before.
18. According to the judgment of the researcher, those who are not suitable for the group, such as poor compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Dose-limiting toxicity
Incidence of treatment related AEs, AEs of special interest and serious adverse events (SAEs). | 2 years
  Assessed by CTCAE V5.0

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  The percentage of subjects with PR or CR assessed by RECIST 1.1.
Overall Survival (OS) | 2 years
  From enrollment to death of patients.
Duration of Response（DOR） | 2 years
  The length of time from the first appearance of a treatment response to the first occurrence of progressive disease or recurrence.
Progression-Free Survival（PFS） | 2 years
  The length of time from enrollment until the time of progression of disease.
Duration of TCR T cells in-vivo persistence | Up to 2 years
  Blood samples were collected to measure persistence of infused HRYZ-T101.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No